CLINICAL TRIAL: NCT07351240
Title: The Quality of Life of Acupuncture Treatment Effect in Patients With Schizophrenia
Brief Title: The Acupuncture Treatment Effect in Patients With Schizophrenia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Calo Psychiatric Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114-051
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mental Health
Keywords: schizophrenia patients; acupuncture; antipsychotic side effects; psychiatric symptoms
MeSH Terms: conditions — Psychological Well-Being | interventions — Acupuncture Therapy

STUDY DESIGN:
Masking Description: Participants will be randomly assigned to either the Neiguan group or the Shenmen group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Effects of Acupuncture on quality of life in schizophrenia (Experimental): It is anticipated that acupuncture will reduce antipsychotic-related side effects, improve psychiatric symptoms in patients with schizophrenia, and subsequently enhance patients' quality of life and happiness.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Both the Neiguan and Shenmen groups will receive acupuncture treatment twice weekly, with each session lasting 30 minutes, for a total of four consecutive weeks. Assessments will be conducted prior to acupuncture intervention and after each acupuncture session.

SUMMARY:
Among various psychiatric disorders, this study focuses specifically on patients with schizophrenia. The aim of this study is to evaluate the therapeutic effects of acupuncture on antipsychotic medication-related side effects and psychiatric symptoms in patients with schizophrenia. This is a single-blind randomized study. Participants will be randomly assigned to one of two groups: Neiguan and Shenmen. Both the Neiguan and Shenmen groups will receive acupuncture treatment twice weekly, with each session lasting 30 minutes, for a total of four consecutive weeks. Assessments will be conducted prior to acupuncture intervention and after each acupuncture session. All assessment data will be collected and analyzed using statistical methods including descriptive statistics, chi-square tests, and t-tests. Generalized Estimating Equations (GEE-I) and multiple linear regression analyses will be applied to examine differences in psychological health, quality of life, and happiness before and after acupuncture intervention. It is anticipated that acupuncture will reduce antipsychotic-related side effects, improve psychiatric symptoms in patients with schizophrenia, and subsequently enhance patients' quality of life and happiness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-5 criteria for at least six months
* Personal and Social Performance Scale score ≥ 50

Exclusion Criteria:

* Severe medical illnesses (e.g., cancer, chronic liver disease, renal failure)
* History of stroke or other causes of hemiplegia
* Severe dermatological disease or limb edema
* High risk of violence or suicide
* Alcohol or substance abuse or dependence
* Severe cognitive impairment
* Pregnancy or breastfeeding
* Severe hepatic, renal, cardiac, pulmonary, or hematological disease
* Major infectious diseases (e.g., HIV infection)
* Refusal to provide informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale | 15 minutes
  assess the anxiety state
Hamilton Depression Scale | 15-20 minutes
  assess the depression state
Short Version of the Udvalg for Kliniske Undersøgelser Side Effect Rating Scale | 5-10 minutes
  assess the psychiatric symptoms

SECONDARY OUTCOMES:
Happiness Scale | 5 minutes
  assess the happiness state

CONTACTS AND LOCATIONS:
Locations (1):
- Calo Psychiatric Center, Pingtung City, Taiwan

IPD SHARING:
Plan to Share IPD: No